CLINICAL TRIAL: NCT00591123
Title: A Phase II Study of Erlotinib and Modified FOLFOX-6 (5-Fluorouracil, Leucovorin and Oxaliplatin) in Previously Untreated Patients With Unresectable or Metastatic Adenocarcinoma of the Esophagus and Gastric Cardia
Brief Title: Study of Erlotinib and Chemotherapy for Unresectable or Metastatic Cancer of the Esophagus and Gastric Cardia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: University of California, Los Angeles (Other); Sanofi (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORI GI-05; BB-IND 77,805 (Other: FDA)
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Results first posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2016-02

CONDITIONS: Unresectable Adenocarcinoma of the Esophagus; Metastatic Adenocarcinoma of the Esophagus; Unresectable Adenocarcinoma of Gastric Cardia; Metastatic Adenocarcinoma of Gastric Cardia
Keywords: Unresectable; Metastatic; Esophagus; Gastric Cardia
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Neoplasm Metastasis | interventions — Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOX, plus 5-FU and Erlotinib (Experimental): single arm
  Interventions: Drug: FOLFOX; Drug: 5-FU; Drug: Erlotinib

INTERVENTIONS:
Drug: FOLFOX — Once every two weeks all patients will receive Oxaliplatin 85 mg/m2 IV, Leucovorin 400 mg/m2 IV and 5-FU 400 mg/m2 IV infusions
  Other Names: Leucovorin Calcium; 5-FU; Oxaliplatin
Drug: 5-FU — 5-FU 2400 mg/m2 IV will be given via pump for 46-48 hours at home.
  Other Names: Fluorouracil
Drug: Erlotinib — All patients will also be given Erlotinib, 100 mg orally daily for the first 4 weeks. Those patients who have not experienced toxicities will increase the dose level to 150 mg daily. Patients who have toxicities will remain at the 100 mg dose level or lower if necessary.

SUMMARY:
In this study, Erlotinib and 5-Fluorouracil (5-FU), Leucovorin and Oxaliplatin (a regimen known also as FOLFOX-6) will be the chemotherapy study drugs. The main purpose of this study is to test the safety and effectiveness of this combination of chemotherapy drugs and to see how they affect your cancer.

Another purpose of this study is to examine samples from your blood and tumor. This research will be done to better understand how subjects respond to treatment. Specifically, researchers will look at the way your genes and proteins respond to drugs like those used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or unresectable adenocarcinoma of the upper gastrointestinal tract that can be measured in at least one dimension according to RECIST criteria by CT or MRI
2. Gastric adenocarcinomas may be included if the primary tumor arises within 5 cm of the anatomic gastro-esophageal junction (distal esophagus) or from the gastric cardia as indicated by either endoscope or imaging.
3. Previously untreated with chemotherapeutic agents for unresectable or metastatic disease.
4. Adjuvant chemotherapy and/or radiotherapy are allowed as long as no oxaliplatin was used in the past 12 months.
5. ECOG performance status 0 or 1
6. Age > 18 years old.
7. Life expectancy greater than 6 months.
8. Peripheral neuropathy: must be < grade 1
9. Absolute neutrophil count > 1,500/mm3
10. Hemoglobin > 9.0 g/dl
11. Platelet count > 100,000/mm3
12. Hepatic Function:

    1. Total Bilirubin < or = to 1.5 x ULN
    2. AST and ALT must be < or = to 3.0 x ULN (< or = to 5.0 x ULN if there is liver metastasis).
13. Creatinine clearance of > 60 ml/min as calculated by the Cockcroft Gault formula. (Ccr = ((140-Age) X Wt (kg))/ (72 X SCr (mg/100ml) for males).

    (Ccr = ((140-Age) X Wt (kg))/ (72 X SCr (mg/100ml) x 0.85 for females)
14. Women of childbearing potential must have a negative pregnancy test by urine or serum testing.
15. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 4 months after the last treatment.
16. Patients must have signed IRB approved informed consent
17. Patients must have the ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. Patients with known hypersensitivity to any components of oxaliplatin, leucovorin, 5-fluorouracil (or other fluoropyrimidines) or erlotinib.
2. Women who are breast-feeding or pregnant.
3. Presence of > Grade 2 neuropathy
4. Patients with prior malignancy other than non-melanoma skin cancer or cervical carcinoma in situ within the past five years
5. Current or prior history of central nervous system or brain metastases
6. Any other medical conditions, which, in the opinion of the investigator, would preclude subjects to participate in the study.
7. Patients who have received chemotherapy, surgery or radiation therapy within 30 days prior to the first dose.
8. INR greater than 3.5 for patients on warfarin
9. Known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev Wainberg, MD, Principal Investigator — University of California, Los Angeles; Fairooz Kabbinavar, MD, Study Director — UCLA - TORI; J Randolph Hecht, MD, Study Chair — University of California, Los Angeles
Locations (2):
- United States (2):
  - Translational Oncology Research International (TORI) Network, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX Plus 5-FU and Erlotinib: FOLFOX and Erlotinib: Once every two weeks all patients will receive Oxaliplatin 85 mg/m2 IV, Leucovorin 400 mg/m2 IV and 5-FU 400 mg/m2 IV infusions, after which 5-FU 2400 mg/m2 IV will be given via pump for 46-48 hours at home. All patients will also be given Erlotinib, 100 mg orally daily for the first 4 weeks. Those patients who have not experienced toxicities will increase the dose level to 150 mg daily. Patients who have toxicities will remain at the 100 mg dose level or lower if necessary.
Period: Overall Study
Arm/Group | FOLFOX Plus 5-FU and Erlotinib
Started | 38
Completed | 38 (38 were analyzed for safety, 33 were included for efficacy.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 50 participants were screened for the study. A total of 12 participants were considered screening failures, 11 did not meet inclusion/exclusion criteria and 1 participant went to Hospice. Thirty eight participants were enrolled.
Arm/Group | FOLFOX Plus 5-FU and Erlotinib
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 38
Eastern Cooperative Group performance status [Number; unit: participants] — ECOG score evaluated during exam by Physician. Runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.)
  2. - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  participants
    0 | 23
    1 | 15
Previous Treatment: Surgery [Number; unit: participants]
  yes | 5
  no | 33
Previous Treatment Chemotherapy [Number; unit: participants]
  Neoadjuvant | 8
  Adjuvant | 30
Previous Chemotherapy Regimens [Number; unit: participants]
  Fluoropyrim/platinum (w/ adjuvant radiation) | 2
  Cisplatin/5-FU based (with neoadjuvant radiation) | 4
  Epirubicin/cisplatin/5-FU | 2
  None | 30
Previous radiation therapy [Number; unit: participants]
  yes | 6
  no | 32
Neoadjuvant vs. Adjuvant Previous Radiation Therapy [Number; unit: participants]
  Neoadjuvant | 4
  Adjuvant | 2
  None | 32
Oesophagus vs. gastro-oesophageal junction [Number; unit: participants]
  Oesophagus | 12
  gastro-oesophageal junction (GEJ) | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Previously-untreated Patients With Unresectable or Metastatic Adenocarcinomas of the Upper Gastrointestinal Tract When Treated With the Combination of 5-fluorouracil, Leucovorin, Oxaliplatin, and Erlotinib.
Description: Per response evaluation criteria in solid tumors criteria (RECIST) for target lesions and assessed by computerized tomography (CT) scan.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 3.5 years
Population: 33 patients who were evaluable for response per protocol
Measure: Number; unit: percent of subjects that had response
Arm/Group | FOLFOX Plus 5-FU and Erlotinib
Number analyzed (Participants) | 33
percent of subjects that had response | 51.5

2. Secondary Outcome: Toxicity of the Combination of FOLFOX, 5-FU, and Erlotinib
Description: Adverse event assessment by investigators and as reported by subjects from time of consent to 30 days after last dose. Up to 3.5 years.
Time Frame: 3.5 years
Population: Number of subjects that experienced Grade 3 and 4 Adverse events associated with FOLFOX/5-FU/Erlotinib therapy
Measure: Number; unit: participants
Arm/Group | FOLFOX Plus 5-FU and Erlotinib
Number analyzed (Participants) | 38
participants
  Diarrhea / dehydration | 9
  Anorexia | 5
  Nausea/Vomiting | 4
  Rash | 3
  Fatigue | 4
  Peripheral neuropathy | 3
  Neutropenia | 5
  Neutropenic Fever | 1
  Hypokalemia | 2
  AST / ALT Elevation | 2

ADVERSE EVENTS:
Time Frame: consent until 30 days post treatment
Description: Systemic adverse event assessment occurred every 14 days through investigator assessment during Treatment Period.
Groups:
- Single Arm: FOLFOX and Erlotinib: Once every two weeks all patients will receive Oxaliplatin 85 mg/m2 IV, Leucovorin 400 mg/m2 IV and 5-FU 400 mg/m2 IV infusions, after which 5-FU 2400 mg/m2 IV will be given via pump for 46-48 hours at home. All patients will also be given Erlotinib, 100 mg orally daily for the first 4 weeks. Those patients who have not experienced toxicities will increase the dose level to 150 mg daily. Patients who have toxicities will remain at the 100 mg dose level or lower if necessary.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 7/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=38)
Neutropenic Fever (Infections and infestations) | 1 (1) — Sepsis associated with neutropenic fever (103°F), hypotension, dehydration, hyponatremia, intermittent gr. 2 diarrhea.
Septic Shock (Infections and infestations) | 1 (1) — Nausea, vomiting, diarrhea, altered mental status, neutropenia with fever, septic shock, renal failure. Participant expired in hospital on 12/26/09.
Malnutrition (General disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Altered Mental State (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Inability to Urinate (Renal and urinary disorders) | 1 (1)
Intractable Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Cranial Hematoma (Injury, poisoning and procedural complications) | 1 (1) — hematoma to head, small acute lacunar infarction.
Finger Infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Elevated International Normalized Ratio (INR) (Blood and lymphatic system disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (2)
diskectomy (Surgical and medical procedures) | 1 (1) — Anterior cervical diskectomy for spinal cord decompression at C5-C6. Diskitis/osteomyelitis at C5-C6. Grade 3 tear of posterior horn of lateral meniscus and a moderate effusion.
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=38)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Alkaline Phosphatase - elevated (Blood and lymphatic system disorders) | 11 (13)
Alopecia (General disorders) | 6 (7)
Alanine Aminotransferase - elevated (Blood and lymphatic system disorders) | 6 (7)
Anemia (Blood and lymphatic system disorders) | 16 (19)
Anorexia (Metabolism and nutrition disorders) | 21 (24)
Aspartate Aminotransferase - elevated (Blood and lymphatic system disorders) | 9 (12)
Blepharitis (Eye disorders) | 1 (1)
Bloating (General disorders) | 5 (6)
Blood in stool (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cachexia (General disorders) | 1 (1)
Cardiac infarction (Cardiac disorders) | 1 (1)
Cerebrovascular accident (CVA) (Vascular disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cold sensitivity (General disorders) | 5 (5)
Cold-like symptoms (General disorders) | 3 (5)
Constipation (General disorders) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cramps - limbs (General disorders) | 3 (3)
Creatinine - elevated (Blood and lymphatic system disorders) | 2 (2)
Dehydration (General disorders) | 14 (15)
Diabetes mellitus (Blood and lymphatic system disorders) | 1 (2)
Diaphoresis (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 28 (53)
Dizziness (General disorders) | 4 (5)
Dry eye (General disorders) | 2 (2)
Dry heaves (General disorders) | 1 (1)
Dry mouth (General disorders) | 4 (4)
Dry Nose (General disorders) | 1 (1)
Dry skin (General disorders) | 9 (10)
Dyspepsia (General disorders) | 3 (5)
Dysphagia (General disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Edema (General disorders) | 7 (12)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (General disorders) | 1 (1)
Facial flushing (General disorders) | 1 (1)
Fatigue (General disorders) | 24 (37)
Fever (General disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (4)
Flu-like syndrome (General disorders) | 1 (1)
Folliculitis (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait-Walking (General disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Glossitis (General disorders) | 1 (1)
Hand and Foot Syndrome (General disorders) | 3 (4)
Heart burn (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemorrhage (GI, gums, nose, upper GI) (General disorders) | 5 (5)
Hemorrhage (nose, oral cavity) (General disorders) | 2 (4)
Hemorrhoid (Gastrointestinal disorders) | 1 (1)
Hiccups (General disorders) | 2 (2)
Hot flashes (Metabolism and nutrition disorders) | 1 (1)
Hyperalbuminemia (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (7)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 9 (11)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 7 (8)
Hypocalcemia (Blood and lymphatic system disorders) | 7 (8)
Hypokalemia (Blood and lymphatic system disorders) | 17 (24)
Hypomagnesia (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 5 (6)
Hypotension (Blood and lymphatic system disorders) | 4 (5)
Hypothermia (General disorders) | 2 (2)
Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Infection (Infections and infestations) | 10 (15) — GI NOS, paronychia, picc line, sinus, skin, skin fungal, ungual, cellulitis, upper airway NOS, urinary tract NOS, J-tube site
Infection (skin, upper airway, pneumonia) (Infections and infestations) | 4 (4)
International Normalized Ratio (INR) - elevated (Blood and lymphatic system disorders) | 2 (2)
Jaundice (Hepatobiliary disorders) | 1 (1)
Joint effusion - Elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
Lactose intolerance (General disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 15 (24)
Lymphopenia (Blood and lymphatic system disorders) | 6 (11)
Mental status (General disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Mood alteration - anxiety (General disorders) | 7 (7)
Mood alteration - depression (General disorders) | 6 (9)
Mucositis - oral cavity (General disorders) | 15 (17)
Myotonia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail Changes (General disorders) | 1 (1)
Nausea (General disorders) | 21 (31)
Neuropathy (Nervous system disorders) | 2 (3)
Neuropathy - motor (Nervous system disorders) | 1 (2)
Neuropathy - sensory (Nervous system disorders) | 22 (38)
Neutropenia (Blood and lymphatic system disorders) | 14 (32)
Neutropenic fever (General disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Obstruction - GI small bowel NOS (Gastrointestinal disorders) | 1 (1)
Ocular - drainage (Eye disorders) | 1 (1)
Ocular - ruptured vessel (Eye disorders) | 1 (1)
Odynophagia (Ear and labyrinth disorders) | 2 (2)
Pain (General disorders) | 29 (48) — abdomen, around J-tube, back, buttock, chest, epigastric, flank, hip, knee, limbs, neck, NOS, rib, shoulder, stomach, throat, right upper quadrant
Pallor (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)
Perforation gastrointestinal tract (Gastrointestinal disorders) | 1 (1)
Performance Status Decrease (General disorders) | 3 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 30 (55) — limbs, chest, scalp, portacath site, facial
Renal failure (Renal and urinary disorders) | 1 (1)
Rhinitis (Ear and labyrinth disorders) | 2 (2)
Rigors-Chills (General disorders) | 3 (3)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
Serum Chloride - Decrease (Blood and lymphatic system disorders) | 2 (2)
Serum Protein - Decreased (Blood and lymphatic system disorders) | 1 (1)
Sinusitis (Ear and labyrinth disorders) | 1 (1)
Hyperpigmentation - portacath site (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) — picc line site
Papule lower extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Papule upper chest (Skin and subcutaneous tissue disorders) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (General disorders) | 1 (1)
Stomatitis (General disorders) | 1 (1)
Sweating (General disorders) | 2 (2)
Syncope (General disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 5 (6)
Taste alteration (General disorders) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombosis-Embolism (Vascular disorders) | 3 (5)
Thrush (Infections and infestations) | 1 (1)
Urinary retention (General disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Voice changes (General disorders) | 1 (1)
Vomiting (General disorders) | 16 (22)
Weakness (General disorders) | 10 (15)
Weight loss (General disorders) | 17 (22)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No